CLINICAL TRIAL: NCT00054184
Title: CT-2103 vs Docetaxel for the Second-Line Treatment of Non-Small Cell Lung Cancer (NSCLC): A Phase III Study
Brief Title: Polyglutamate Paclitaxel Compared With Docetaxel in Treating Patients With Progressive Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTI-PGT302; CDR0000269907 (Registry Identifier: PDQ (Physician Data Query)); CWRU-CTI-1503
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IV non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; paclitaxel poliglumex

ARMS (1):
- Study drug (Experimental)
  Interventions: Drug: docetaxel; Drug: paclitaxel poliglumex

INTERVENTIONS:
Drug: docetaxel
Drug: paclitaxel poliglumex

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether polyglutamate paclitaxel is more effective than docetaxel in treating non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of polyglutamate paclitaxel with that of docetaxel in treating patients who have progressive non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of polyglutamate paclitaxel (CT-2103) vs docetaxel as second-line therapy, in terms of duration of overall survival, in patients with progressive non-small cell lung cancer.
* Compare the safety and toxicity of these regimens in these patients.
* Compare the disease control (stable disease maintained for at least 12 weeks, partial response, or complete response) and progression-free survival of patients treated with these regimens.
* Compare the improvement in lung cancer symptoms in patients treated with these regimens.
* Compare the frequency of grade 3 and 4 neurotoxicity, edema, alopecia, and side effects related to corticosteroids in patients treated with these regimens.
* Determine the percentage of patients who receive at least 4 courses of study treatment.
* Compare the response rate in patients with measurable disease treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to stage (IV vs other), performance status (0 or 1 vs 2), start of front-line chemotherapy from randomization (less than 16 weeks vs at least 16 weeks), gender, and prior taxane therapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive polyglutamate paclitaxel (CT-2103) IV over 10 minutes on day 1.
* Arm II: Patients receive docetaxel IV over 1 hour on day 1. In both arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at 3 weeks and then every 8 weeks thereafter.

PROJECTED ACCRUAL: A total of 840 patients (420 per treatment arm) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer (NSCLC)
* Documented clinical or radiologic disease progression on or after initial systemic therapy

  * Must have received 1 prior platinum-based systemic therapy for NSCLC
* Measurable or nonmeasurable disease
* No evidence of small cell carcinoma, carcinoid, or mixed small cell/non-small cell histology
* Brain metastases allowed provided patient received prior standard antitumor therapy for CNS metastases (e.g., whole brain radiotherapy, stereotactic radioablation, or surgery) and the following conditions are met:

  * No prior systemic chemotherapy as a radiosensitizer combined with radiotherapy
  * Obtained stable neurologic function at least 2 weeks before study entry
  * Off steroid therapy or on a tapering regimen
  * Recovered from prior therapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Al least 16 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN
* AST or ALT no greater than 1.5 times ULN

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* No unstable angina
* No myocardial infarction within the past 6 months
* No evidence of cardiac conduction abnormalities (e.g., bundle branch block or heart block) unless cardiac status stable for the past 6 months

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No evidence of unstable neurological symptoms in the past 4 weeks (2 weeks for neurological symptoms due to brain metastases)
* No intolerance to excipients of polyglutamate paclitaxel (e.g., poly-L-glutamic acid, poloxamer 188, dibasic sodium phosphate, or monobasic sodium hydroxide)
* No other unstable medical conditions
* No clinically significant active infection
* No neuropathy greater than grade 1
* No other concurrent primary malignancy except carcinoma in situ or nonmelanoma skin cancer
* No circumstance that would preclude study completion or follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No prior polyglutamate paclitaxel
* No prior docetaxel

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* See Disease Characteristics
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* Recovered from prior major surgery

Other

* Recovered from prior therapy
* More than 2 weeks since prior treatment for NSCLC
* More than 4 weeks since prior investigational drugs
* No other concurrent investigational drugs
* No other concurrent systemic antitumor therapy
* No concurrent amifostine
* Concurrent bisphosphonates allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2003-01 (Actual); Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Saftey | Baseline to end of treatment

SECONDARY OUTCOMES:
Efficacy | Basline to EOS

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Garrison, Study Chair — PPD, Incorporated
Locations (35):
- United States (35):
  - Clinical Research Consultants, Incorporated, Hoover, Alabama
  - Arizona Clinical Research Center, Tucson, Arizona
  - Highlands Oncology Group - Springdale, Springdale, Arkansas
  - Pacific Cancer Medical Center, Incorporated, Anaheim, California
  - Synergy Hematology/Oncology Medical Associates, Encino, California
  - California Cancer Care, Inc., Greenbrae, California
  - California Hematology/Oncology Medical Group, Torrance, California
  - Northwest Oncology and Hematology Associates, Coral Springs, Florida
  - Florida Oncology Associates, Jacksonville, Florida
  - Hematology Oncology Associates of theTreasure Coast - Port St. Lucie, Port Saint Lucie, Florida
  - Suburban Hematology-Oncology, Snellville, Georgia
  - Gross Point Medical Center, Skokie, Illinois
  - Western Kentucky Hematology/Oncology Group, Paducah, Kentucky
  - Kentucky Cancer Clinic, Pikeville, Kentucky
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - Montana Cancer Specialists, Missoula, Montana
  - Las Vegas Cancer Center, Las Vegas, Nevada
  - Howell Township, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - New Mexico Oncology-Hematology Consultants, Limited, Albuquerque, New Mexico
  - Queens Medical Associates, PC, Fresh Meadows, New York
  - Piedmont Oncology Specialist, II, PLLC, Monroe, North Carolina
  - Odyssey Research Services, Bismarck, North Dakota
  - Gabrail Cancer Center - Canton Office, Canton, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - Charleston Hematology-Oncology, P.A., Charleston, South Carolina
  - Tri County Oncology Associates, Rock Hill, South Carolina
  - Santee Hematology Oncology, Sumter, South Carolina
  - Family Cancer Center, Collierville, Tennessee
  - Southwest Regional Cancer Center, Austin, Texas
  - Richardson, Texas
  - Danville Hematology and Oncology, Incorporated, Danville, Virginia
  - Virginia Oncology Care P.C., Richlands, Virginia
  - Western Washington Medical Group, Everett, Washington